CLINICAL TRIAL: NCT00036751
Title: A Phase II Trial Of STI571 For The Treatment Of Platinum And Taxane Refractory Stage III And IV Epithelial Ovarian Cancer And Primary Peritoneal Cancer
Brief Title: Imatinib Mesylate in Treating Patients With Stage III or Stage IV Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02463; SWOG-S0211; U10CA032102 (NIH); CDR0000069319 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have stage III or stage IV ovarian epithelial or primary peritoneal cancer that has not responded to previous treatment. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rates (confirmed, complete, and partial) in patients with platinum- and taxane-refractory stage III or IV ovarian epithelial or primary peritoneal cancer treated with imatinib mesylate.

II. Determine the toxicity of this drug in these patients. III. Correlate, preliminarily, CD117 and platelet-derived growth factor receptor expression levels with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial carcinoma of the ovary or primary peritoneal serous papillary carcinoma

  * No mixed Mullerian tumors
  * No borderline ovarian tumors
* Stage III or IV disease at time of diagnosis by surgical staging
* Expression of KIT (CD117) and/or platelet-derived growth factor receptor by immunohistochemistry
* Relapsed within 6 months after completion of or progressed while receiving prior frontline chemotherapy with a platinum (cisplatin or carboplatin) and a taxane(paclitaxel or docetaxel) administered concurrently or sequentially
* Measurable disease
* Performance status - Zubrod 0-1
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No New York Heart Association class III or IV heart disease (e.g., congestive heart failure or myocardial infarction within the past 2 months)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other adequately treated stage I or II cancer in complete remission
* At least 28 days since prior biologic therapy
* No concurrent anticancer biologic therapy
* No concurrent cytokines (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* At least 28 days since prior chemotherapy
* No more than 3 prior chemotherapy regimens in addition to frontline chemotherapy

  * Retreatment with a platinum agent or with the same taxane as in the frontline regimen is not counted as an additional regimen
* No concurrent chemotherapy
* Prior hormonal therapy allowed
* Recovered from prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy
* Prior surgical debulking allowed for relapsed disease if measurable disease remains after surgery
* At least 14 days since prior major surgery
* Recovered from all prior surgery
* At least 28 days since prior investigational drugs
* No concurrent therapeutic doses of warfarin for anticoagulation (heparin or mini-dose warfarin (1 mg/day) allowed)
* No other concurrent anticancer agents
* No other concurrent investigational drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-04; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial confirmed response) | Up to 3 years

SECONDARY OUTCOMES:
Toxicity as assessed by NCI Common Toxicity Criteria version 2.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Alberts, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group (SWOG) Research Base, San Antonio, Texas, United States